CLINICAL TRIAL: NCT02089256
Title: Effect of Repeated Administration of Liraglutide on Insulinogenic Indices
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Vallo Volke, Professor, University of Tartu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LI20/1101
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Healthy
MeSH Terms: interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Liraglutide (Experimental): Liraglutide 0.6 mg/day subcutaneously.
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — Graded glucose infusion test (GGIT)will be performed on baseline. 1 week later treatment with liraglutide 0.6mg/day (injected between 21.00-23.00) will be initiated.
  GGIT will be repeated 12 hours after first injection and after 21 days on-treatment (12 hours after last injection).
  Other Names: Victoza

SUMMARY:
The study investigates the effect of glucagon-like peptide receptor 1 agonist, liraglutide, on insulin secretion. Study hypothesis: the effect of liraglutide on insulin release may change after repeated administration. The effect of liraglutide on insulin release will be tested using graded glucose infusion test (GGIT) in healthy volunteers. GGIT will be performed without medication and repeated 12 hours after first dose of liraglutide and after 3 weeks of treatment with liraglutide.

ELIGIBILITY:
Inclusion Criteria:

* Weight 50-100 kg

Exclusion Criteria:

* Chronic disease
* Concomitant drug use
* Pregnancy or lactation
* Fasting glucose >6 mmol/L.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in the glucose-sensitivity of the beta cells | baseline, first dose, after 3-weeks on treatment
  Graded glucose infusion test will be used to create insulin secretion rate- plasma glucose curve. The primary outcome is the change of the slope of the curve from baseline after acute administration of liraglutide compared to the repeated administration (after 3-weeks of treatment).

SECONDARY OUTCOMES:
Effects on adrenal hormones | baseline, acute administration, 3 weeks
  change in ACTH/cortisol levels and renin / aldosterone levels after acute and repeated administration of liraglutide.

CONTACTS AND LOCATIONS:
Overall Officials: Vallo Volke, MD, Principal Investigator — University of Tartu
Locations (1):
- Tartu University Hospital, Tartu, Estonia

REFERENCES:
- [Derived] Heinla K, Vasar E, Reppo I, Sedman T, Volke V. GLP-1 Receptor Agonists Induce Growth Hormone Secretion in Healthy Volunteers. Diabetes Ther. 2023 Apr;14(4):777-786. doi: 10.1007/s13300-023-01381-w. Epub 2023 Feb 17. PMID 36800161
- [Derived] Sedman T, Vasar E, Volke V. Tolerance Does Not Develop Toward Liraglutide's Glucose-Lowering Effect. J Clin Endocrinol Metab. 2017 Jul 1;102(7):2335-2339. doi: 10.1210/jc.2017-00199. PMID 28379427
- [Derived] Sedman T, Heinla K, Vasar E, Volke V. Liraglutide Treatment May Affect Renin and Aldosterone Release. Horm Metab Res. 2017 Jan;49(1):5-9. doi: 10.1055/s-0042-109065. Epub 2016 Jun 14. PMID 27300475